CLINICAL TRIAL: NCT07220187
Title: A Randomized Phase III Study of Pirtobrutinib Plus R-CHOP vs. R-CHOP for Participants With Previously Untreated Richter Transformation (PIRAMID)
Brief Title: Adding Pirtobrutinib to the Usual Treatment for People With Newly Diagnosed Richter Transformation, The PIRAMID Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2504; NCI-2025-06717 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2504 (Other: SWOG); S2504 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2025-10-06; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Richter Syndrome; Transformed Chronic Lymphocytic Leukemia to Diffuse Large B-Cell Lymphoma; Transformed Small Lymphocytic Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: interventions — Specimen Handling; Cyclophosphamide; Doxorubicin; pirtobrutinib; Magnetic Resonance Spectroscopy; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Hyaluronoglucosaminidase; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (pirtobrutinib and R-CHOP) (Experimental): Patients receive pirtobrutinib PO QD on days 1-21 of each cycle, rituximab IV or rituximab hyaluronidase SC (starting with cycle 2), cyclophosphamide IV on day 1 of each cycle, doxorubicin IV on day 1 of each cycle, vincristine IV on day 1 of each cycle, and prednisone PO QD on days 1-5 of each cycle. Cycles repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After completion of cycle 6, patients continue to receive pirtobrutinib PO QD on days 1-21 of each cycle for up to 5 years in the absence of disease progression or unacceptable toxicity. Patients with progressive disease or symptomatic deterioration may receive 1 additional cycle as long as the participant is continuing to clinically benefit from treatment in the opinion of the treating investigator. Patients undergo echocardiography or MUGA scan and buccal swab collection during screening, as well as CT scan and/or PET/CT, and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Pirtobrutinib; Procedure: Positron Emission Tomography; Drug: Prednisone; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human; Other: Survey Administration; Drug: Vincristine
- Arm II (R-CHOP) (Active Comparator): Patients receive rituximab IV or rituximab hyaluronidase SC (starting with cycle 2), cyclophosphamide IV on day 1 of each cycle, doxorubicin IV on day 1 of each cycle, vincristine IV on day 1 of each cycle, and prednisone PO QD on days 1-5 of each cycle. Cycles repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography or MUGA scan and buccal swab collection during screening, as well as CT scan and/or PET, and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Drug: Prednisone; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human; Other: Survey Administration; Drug: Vincristine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and buccal swab sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan and/or PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Pirtobrutinib — Given PO
  Other Names: 5-Amino-3-(4-((5-fluoro-2-methoxybenzamido)methyl)phenyl)-1-((2S)-1,1,1-trifluoropropan-2-yl)-1h-pyrazole-4-carboxamide; BTK Inhibitor LOXO-305; Jaypirca; LOXO 305; LOXO-305; LOXO305; LY3527727
  Arms: Arm I (pirtobrutinib and R-CHOP)
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Biological: Rituximab and Hyaluronidase Human — Given SC
  Other Names: Rituxan Hycela; Rituximab Plus Hyaluronidase; Rituximab/Hyaluronidase; Rituximab/Hyaluronidase Human
Other: Survey Administration — Ancillary studies
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This phase III trial compares the effect of adding pirtobrutinib to the usual treatment with rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone (R-CHOP) to R-CHOP alone for the treatment of Richter transformation, which is when chronic lymphocytic leukemia or small lymphocytic lymphoma turns into large B-cell lymphoma, a more aggressive (faster-growing) form of lymphoma. Pirtobrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill cancer cells. It may also lower the body's immune response. Doxorubicin is in a class of medications called anthracyclines. Doxorubicin damages the cell's DNA and may kill cancer cells. It also blocks a certain enzyme needed for cell division and DNA repair. Vincristine is in a class of medications called vinca alkaloids. It works by stopping cancer cells from growing and dividing and may kill them. Prednisone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Adding pirtobrutinib to R-CHOP may kill more cancer cells than R-CHOP alone in patients with Richter transformation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. In participants aged 74 and younger, to evaluate the safety of the addition of pirtobrutinib to R-CHOP before initiating randomization in participants with untreated Richter Transformation to large B-cell lymphoma (LBCL). (Safety run-in) II. In participants aged 75 and older, to evaluate the safety of the addition of pirtobrutinib to R-mini-CHOP before initiating randomization in this patient population. (Safety run-in) III. To evaluate whether the addition of pirtobrutinib to R-CHOP improves investigator-assessed progression-free survival (PFS) compared to R-CHOP alone in this patient population. (Randomized comparison) IV. If investigator-assessed PFS is improved with the addition of pirtobrutinib, then to evaluate whether the addition of pirtobrutinib improves overall survival (OS) in this patient population. (Randomized comparison-hierarchical testing)

TRANSLATIONAL MEDICINE PRIMARY OBJECTIVE:

I. To evaluate the association between high-risk Richter-associated mutations (presence vs. absence of at least one of: TP53, CDK2NA, or MYC pathway alterations as assessed by targeted next generation sequencing (NGS) panel and whole exome sequencing of baseline tumor tissue) and overall survival (OS) within treatment arms in this patient population.

SECONDARY OBJECTIVES:

I. To estimate and compare the rate of investigator-assessed complete response (CR) after treatment between the randomized arms.

II. To estimate the frequency and severity of adverse events in both arms.

TRANSLATIONAL MEDICINE SECONDARY OBJECTIVES:

I. To evaluate the association between high-risk Richter-associated mutations and overall response rate (ORR [complete and partial response], PFS and complete response [CR]) across treatment arms in this patient population.

II. To descriptively report the interaction between high-risk Richter-associated mutations and randomized arm and the outcomes CR, ORR, PFS, and OS.

III. To descriptively report the mutational landscape (as assessed by targeted NGS panel and whole exome sequencing of baseline tumor tissue and at the time of progression) in this patient population.

IV. In mutations present in at least 5 patients, to descriptively report CR, ORR, PFS, and OS by mutation status across treatment arms.

V. To evaluate associations between minimal residual disease (MRD) status (as assessed by circulating tumor deoxyribonucleic acid [ctDNA]) and OS and PFS.

VI. To evaluate associations between clonal relatedness and OS and PFS across treatment arms.

ADDITIONAL OBJECTIVES:

I. To compare OS of participants receiving stem cell transplant versus those who did not receive transplant.

II. To compare the OS of participants receiving chimeric antigen receptor t cell (CAR-T) therapy versus those who did not receive CAR-T therapy.

III. To evaluate the association between Bruton Tyrosine Kinase (BTK) resistance mutations on clinical outcomes (PFS and OS).

IV. To evaluate the association of clonal relatedness between chronic lymphocytic leukemia (CLL) and LBCL and clinical outcomes (PFS and OS).

PATIENT-REPORTED OUTCOMES OBJECTIVE:

I. To compare participant-reported symptoms (PROs) between arms as measured by PRO-Common Terminology Criteria for Adverse Events (CTCAE) items and the Functional Assessment of Chronic Illness Therapy (FACIT) single-item GP5 question.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive pirtobrutinib orally (PO) once daily (QD) on days 1-21 of each cycle, rituximab intravenously (IV) or rituximab and hyaluronidase human (rituximab hyaluronidase) subcutaneously (SC) (starting with cycle 2), cyclophosphamide IV on day 1 of each cycle, doxorubicin IV on day 1 of each cycle, vincristine IV on day 1 of each cycle, and prednisone PO QD on days 1-5 of each cycle. Cycles repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After completion of cycle 6, patients continue to receive pirtobrutinib PO QD on days 1-21 of each cycle for up to 5 years in the absence of disease progression or unacceptable toxicity. Patients with progressive disease or symptomatic deterioration may receive 1 additional cycle as long as the participant is continuing to clinically benefit from treatment in the opinion of the treating investigator. Patients undergo echocardiography or multigated acquisition (MUGA) scan and buccal swab collection during screening, as well as computed tomography (CT) scan and/or positron emission tomography (PET)/CT, and blood sample collection throughout the study.

ARM 2: Patients receive rituximab IV or rituximab hyaluronidase SC (starting with cycle 2), cyclophosphamide IV on day 1 of each cycle, doxorubicin IV on day 1 of each cycle, vincristine IV on day 1 of each cycle, and prednisone PO QD on days 1-5 of each cycle. Cycles repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography or MUGA scan and buccal swab collection during screening, as well as CT scan and/or PET, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up periodically for until 7 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been diagnosed with Richter Transformation (RT) (CLL/small lymphocytic lymphoma [SLL] to LBCL)

  * Participants must have histologically or cytologically confirmed LBCL
* Participants must have measurable disease determined by PET/CT or hematopathology (by morphology or flow cytometry) assessment within 42 days prior to registration
* Participants must have staging PET/CT imaging performed within 42 days prior to registration
* Participants are allowed prior treatments for CLL/SLL or its complications (autoimmune hemolytic anemia [AIHA], immune thrombocytopenic purpura [ITP]), with the exception of pirtobrutinib
* Participants must not have prior treatment for Richter transformation except for corticosteroids up to equivalent dose of prednisone 700 mg total for less than 7 days for disease control. Treatment for CLL/SLL with CLL/SLL directed drugs (including BTK inhibitors with the exception of pirtobrutinib) after the Richter transformation diagnosis is allowed for the purpose of disease control. CLL targeted therapies must be stopped within 3 days before initiation of therapy on protocol. Chemotherapy or anti-CD20 monoclonal antibody therapy must be stopped within 2 weeks before initiation of therapy on protocol
* Participants must not have contraindication for receiving anthracycline. Participants must not have received more than a cumulative dose of 100mg/m^2 in those participants who will receive R-CHOP or not more than 250 mg/m^2 in those participants who will receive R-mini-CHOP of prior doxorubicin (or equivalent dose of another anthracycline, such as epirubicin) therapy (at any time prior to registration)
* Patients requiring strong CYP3A inducers are not eligible and can only be enrolled if

  * an alternative treatment to the strong CYP3A inducer is available for them and
  * the last dose of the strong CYP3A inducer is administered at least 7 days before initiation of pirtobrutinib for patients in safety run-in and arm 1
* Participant must be ≥ 18 years old at the time of registration
* Participant must have Eastern Cooperative Oncology Group (ECOG)/Zubrod Performance Status of 0-2
* Participant must have a complete medical history and physical exam within 28 days prior to registration
* Absolute neutrophil count (ANC) ≥ 0.75 x 10^3/µL or ≥ 0.50 x 10^3/µL in participants with suspected marrow involvement considered to impair hematopoiesis (within 28 days prior to registration)
* Platelets ≥ 50 x 10^3/µL or ≥ 30 x 10^3/µL in participants with suspected marrow involvement considered to impair hematopoiesis (within 28 days prior to registration)
* Hemoglobin ≥ 8 g/dL (≥ 80 g/L) or ≥ 6 g/dL in participants with suspected bone marrow involvement considered to impair hematopoiesis (within 28 days prior to registration)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) or ≤ 3 x ULN with documented liver involvement and/or Gilbert's disease (within 28 days prior to registration)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 3 × institutional ULN or ≤ 5 ULN with documented liver involvement (within 28 days prior to registration)
* Participants must have a calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to registration. For the Cockcroft-Gault formula for calculated creatinine clearance, see the tools on the CRA Workbench https://txwb.crab.org/TXWB/Tools.aspx
* Participants must have a left ventricular ejection fraction (LVEF) ≥ 45% as measured by echocardiogram or radionuclide (MUGA) ventriculography within 56 days prior to registration
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Participants' HIV-directed therapy cannot have known interactions with pirtobrutinib
* Participants with a known history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to registration
* Participants with a known history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to registration
* Participants must be able to swallow and retain oral medications and have no known gastrointestinal disorders likely to interfere with absorption of oral medications
* Participants must not have a prior or concurrent malignancy in addition to CLL/SLL and Richter transformation whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not have had major surgery within 28 days prior to registration
* Participants must not have experienced a major bleeding event or grade ≥ 3 arrhythmia on prior treatment with a BTK inhibitor.

  * NOTE: Major bleeding is defined as bleeding having one or more of the following features: potentially life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the hemoglobin level of at least 2g per deciliter; or bleeding in a critical area or organ (e.g., retroperitoneal, intraarticular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome
* Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must be offered the opportunity to participate in specimen banking
* Participants must agree to have blood and lymphatic tissue specimens submitted for the integrated translational medicine study
* For randomized participants only: Participants who can complete PRO-CTCAE and FACIT GP5 questionnaires forms in English or Spanish must be offered the opportunity to participate in the patient-reported outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-05-02 (Estimated); Primary Completion 2035-10-01 (Estimated); Study Completion 2036-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 7 years
  Progression free survival: is measured from date of randomization to the first of progression or death from any cause. Participants last known to be alive without progression will be censored at the date of last contact.
Overall free survival | Up to 7 years
  Overall free survival: is measured from date of randomization date of death from any cause. Participants last known to be alive will be censored at the date of last contact.

SECONDARY OUTCOMES:
Overall Response | Up to 7 years
  Will estimate outcomes (CR, ORR, MRD) for each arm as proportions with binomial confidence intervals. Proportions will be compared between arms using Fisher's exact test.
Complete Remission | Up to 7 years
  Complete disappearance of all measurable and non-measurable disease.
Incidence of adverse events | Up to 7 years
  Number of patients with grade 3 through 5 adverse events that are related (possibly, probably, definitely) to protocol therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mazyar Shadman, Principal Investigator — SWOG Cancer Research Network